CLINICAL TRIAL: NCT01237184
Title: Comparison of Initial Implant Stability of Posterior Maxillary Implants With Bicortical Fixation to Implants Engaging Only the Alveolar Crest
Brief Title: Initial Stability of Posterior Maxillary Implants With Bicortical Fixation
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: 1003M78573; D-2010-021 (Other: Astra Tech)
Record Dates: First submitted 2010-11-01; First posted 2010-11-09 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Tooth Loss
Keywords: initial dental implant stability; maxillary sinus proximity; bicortical fixation
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- biocortical fixation: Bi-cortically fixed implants intentionally engaging sinus floor beyond up to 1-2mm without graft but using stopper drill and self-threading concept
- unicortical fixation: Short implants placed in proximity of the sinus without sinus floor involvement
- indirect sinus lift: implants engaging both crest and sinus floor but with green stick fracture

SUMMARY:
The primary purpose of this study is to

1. determine whether dental implant engaging both the alveolar crest cortical bone and sinus floor using vertical stopper drill and self-threading concept (bi-cortical fixation) increases initial implant stability compared to the short implants engaging only alveolar crest cortical bone (uni-cortical fixation) and/or ones engaging both crest and sinus floor but with green stick fracture (indirect sinus lift technique),
2. study whether different surgical techniques, residual bone height, bone density, and length and width of the implants used affect initial implant stability in posterior maxilla. In addition, this study will continue to
3. compare secondary implant stability of implants fixed bi-cortically, uni-cortically and with indirect sinus lift technique at 2nd stage surgery/6 month healing and 1 year follow-up from the restoration and
4. measure amount of endo-sinus bone formation from the 1- year follow up CT (computer tomogram) scan and evaluate safety and potential post-operative complications of bi-cortical fixation and indirect sinus lift technique reported throughout the follow up periods.

DETAILED DESCRIPTION:
The clinical trial will evaluate initial implant stability as a primary outcome measured by resonance frequency analysis (RFA) employing dental implants surgically placed in posterior maxillary bone by engaging alveolar crest and the sinus floor using vertical stopper drill and self-threading concept (bi-cortical fixation), engaging only the alveolar crest (uni-cortical fixation), and engaging alveolar crest and the sinus floor using indirect sinus lift technique (indirect sinus lift technique). The surgical procedures compared in this experiment include 3 groups:

* Group 1 (15 implants) Short implants placed in proximity of the sinus without sinus floor involvement (unicortical fixation)
* Group 2 (15 implants) Implants placed using indirect sinus lift technique (indirect sinus lift technique)
* Group 3 (15 implants) Bi-cortically fixed implants intentionally engaging sinus floor beyond up to 1-2mm without graft but using stopper drill and self-threading concept (bi-cortical fixation)

ELIGIBILITY:
Inclusion Criteria:

* Eligible volunteers must be at least 18 years old, partially edentulous in maxillary posterior region with 7-11 mm residual bone height under the sinus floor and be indicated for CBCT scan for diagnosis and treatment planning, and of a medical risk of ASA I or II classification to participate.

Exclusion Criteria:

* Patients with bone pathology, sinus infection, and who are pregnant will be excluded. Implants requiring tapping, site of an implant replacement, and implant with dehiscence and/or fenestration will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible volunteers must be at least 18 years old, partially edentulous in maxillary posterior region with 7-11 mm residual bone height under the sinus floor and be indicated for CBCT scan for diagnosis and treatment planning, and of a medical risk of ASA I or II classification to participate. Patients with bone pathology, sinus infection, and who are pregnant will be excluded.
  Implants requiring tapping, site of an implant replacement, and implant with dehiscence and/or fenestration will be excluded.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
initial implant stability | measued immediately after each dental implant is placed in patient's mouth.
  The investigators expect the recruitments and implant placement surgeries for 45 implants will take a year so initial implant stability of each one of 45 implants will be measured over the 1 year period.

CONTACTS AND LOCATIONS:
Overall Officials: Wook-Jin Seong, DDS, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Dental school clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No